CLINICAL TRIAL: NCT03946189
Title: Comparison of the PaO2/FiO2 Ratio to Other Oxygenation Indexes for the Classification of Severity of Acute Respiratory Distress Syndrome
Status: Completed | Type: Observational
Sponsor: American University of Beirut Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: BIO-2018-0033
Record Dates: First submitted 2019-05-09; First posted 2019-05-10 (Actual); Last update posted 2019-05-10 (Actual); Status verified 2019-05

CONDITIONS: Acute Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- P/F less than 100: Patients receiving mechanical ventilation with paO2/FiO2 less than 100
  Interventions: Diagnostic Test: Obtaining arterial blood gases
- P/F between 100 and 200: Patients receiving mechanical ventilation with paO2/FiO2 between 100 and 200
  Interventions: Diagnostic Test: Obtaining arterial blood gases
- P/F between 200-300: Patients receiving mechanical ventilation with paO2/FiO2 between 200 and 300
  Interventions: Diagnostic Test: Obtaining arterial blood gases

INTERVENTIONS:
Diagnostic Test: Obtaining arterial blood gases — Obtaining arterial blood sample
  Other Names: No other intervention

SUMMARY:
In mechanically ventilated patients the PaO2/FiO2 ratio might not be the best reflection of the severity of ARDS. It does not incorporate variables and settings used during mechanical ventilatory support such as the positive end expiratory pressure (PEEP), inspiratory time to expiratory time ratio (Ti:Te), and the peak alveolar pressure (Palv). The aim is to identify a new oxygenation index for stratification of severity of ARDS

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving mechanical ventilation in the Intensive Care Unit.
* Patients in whom the managing medical team requested an arterial blood gas (ABG) analysis.

Exclusion Criteria:

* Patients in whom arterial blood gas could not be obtained or not ordered.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients of both gender and greater than 18 years old receiving mechanical ventilation in the ICU
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2018-03-14 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
New oxygenation index | Immediate
  Oxygenation index that incorporates ventilator parameters

CONTACTS AND LOCATIONS:
Locations (1):
- American University of Beirut, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] El-Khatib MF, Bouakl IJ, Ayoub CM, Chatburn RL, Farhat H, Msheik M, Fakih MH, Hallal AH. Comparison of the Oxygenation Factor and the Oxygenation Ratio in Subjects With ARDS. Respir Care. 2020 Dec;65(12):1874-1882. doi: 10.4187/respcare.07669. Epub 2020 Jul 21. PMID 32694182